CLINICAL TRIAL: NCT05000801
Title: Safety and Feasibility Study of Dendritic Cell (DC) Vaccination Expressing WT1/hTERT/Survivin in AML Patients With Minimal Residual Disease (MRD)
Brief Title: Clinical Study of DC-AML Cells in the Treatment of Acute Myeloid Leukemia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 307-DC-1911
Record Dates: First submitted 2021-07-13; First posted 2021-08-11 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — lentiviral minigene vaccine of COVID-19 coronavirus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DC vaccine (Experimental): Vaccination with autologous or HLA-matched donors' WT1/TERT/survivin loaded DCs plus follow-up care.
  Interventions: Biological: DC vaccine

INTERVENTIONS:
Biological: DC vaccine — Autologous/or HLA-matched donors' DCs loaded with WT1/TERT/survivin

SUMMARY:
The primary aim of this innovative immunotherapy using WT1/hTERT/Survivin-loaded DCs is to determine whether this novel DC vaccination is safe and can significantly prevent clinical relapse and increase survival of acute myeloid leukemia (AML) patients by eradicating minimal residual disease, while maintaining its safety profile in this phase I trial.

DETAILED DESCRIPTION:
we will conduct a single-arm phase I clinical study in 20 patients with acute myeloid leukemia (AML) at the stage of minimal residual disease (MRD) following standard chemotherapy, and these patients are not the subjects of stem cell transplantation. Adult patients between18 and 70 years old with AML who have entered morphological remission after induction, consolidation or intensive chemotherapy with molecular signature of increased WT1 molecule levels and pathological characteristics of bone marrow biopsy, together with fulfilling all other eligibility criteria, will be vaccinated with dendritic cells loaded with tri-antigens (WT1/TERT/survivin) in the absence of any additional therapeutic measurements. The primary aim of this innovative immunotherapy study is to determine whether the anti-leukemic effects seen in our preclinical study can be confirmed in patients and whether such DC vaccination can significantly prevent relapse and increase survival of AML patients by eradicating minimal residual disease. Patients will be recruited at 307 Hospital in Beijing. Recruitment will start in the second half of 2021 and will last for two years or until 20 safety and efficacy-evaluable AML patients are included. This is a single-arm trial. The patients who present MRD after complete chemotherapy will receive a conditioning regimen of cyclophosphamide, followed by six infusions of autologous or HLA-matched donor-derived DCs loaded with tri-antigens including WT1/TERT/survivin. The dendritic cell therapy product will be administered in the stem cell transplantation center at 307 Hospital headed by Dr. Liang-Ding Hu. After inclusion of 20 safety/feasibility-evaluable patients, relapse rate, relapse-free survival and overall survival analysis will be performed. Tumor marker levels and immune signature molecules will also be monitored at molecular and immunological levels, and general and disease-specific quality of life will be evaluated using quality of life questionnaires at various time points.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute myeloid leukemia (AML) according to the 2008 criteria of the World Health Organization (WHO).
* Patients completed induction and consolidation chemotherapy and have achieved complete remission (CR) by bone marrow biopsy criteria but with persistent MRD (defined by upregulated WT1 level and less than 5% of blast cells in bone marrow biopsy) and are not eligible for stem cell transplant
* Patients have MRD molecular relapse (defined by upregulated WT1 level and less than 5% of blast cells in bone marrow biopsy) after achieved CR following induction and consolidation chemotherapy.
* Patients with molecular relapse (define by upregulated WT1 level and less than 5% of blast cells in bone marrow biopsy) after allogeneic stem cell transplant
* Leukemic cells express at least one of the following antigens: WT1, hTERT or survivin detected by qRT-PCR and/or flow cytometry or immunohistochemistry
* Karnofsky PS ≥60% or ECOG PS≤2.
* Patients must have organ and marrow function as defined below:

  * leukocytes >=3,000/mcL
  * absolute neutrophil count >=1,500/mcL
  * platelets >=100,000/mcL
  * hemoglobin >=9.0 g/dL
  * total bilirubin within normal institutional limits except in patients with Gilberts Syndrome who must have a total bilirubin < 3.0 mg/dL
  * AST(SGOT)/ALT(SGPT) Serum ALT/AST < 2.5X ULN
  * creatinine clearance Calculated creatinine clearance (CrCl) >=50 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal (by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation)
  * Adequate cardiac function: LVEF ≥50% by MUGA
* Ability of subject to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participation in any other interventional clinical trial during the study period.
* History or concomitant presence of any other malignancy, except for any other effectively treated malignancy that has been in remission for >5 years or that is highly likely to be cured at the time of enrollment.
* Patients with a second invasive malignancy requiring treatment within the last 2 years are not eligible.
* Patients with any form of systemic immunodeficiency, including AIDS or primary immunodeficiency such as Severe Combined Immunodeficiency Disease, are ineligible. The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the treatment.
* Active hepatitis B, C infection
* Patients on immunosuppressive drugs including corticosteroids.
* Patients with autoimmune diseases such as Crohn s disease, ulcerative colitis, rheumatoid arthritis, autoimmune hepatitis, autoimmune pancreatitis, or systemic lupus erythematosus.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations at the time of treatment that would limit compliance with study requirements.
* Allergic to human albumin or IL-2. History of severe allergic reactions attributed to compounds of similar chemical or biologic composition to agents used in study.
* Pregnant or breast-feeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
the Incidence of Treatment Adverse Events | through study completion,an average of 3 years
  To determine the safety of autologous/or HLA-matched DCs loaded with WT1/TERT/Survivin. The primary objective of this single-arm phase I clinical study is to determine the safety and feasibility of WT1/TERT/survivin-targeted DC vaccination in adult AML patients with MRD at very high risk of relapse.

SECONDARY OUTCOMES:
OS | through study completion,an average of 3 years
  Overall survival
Complete MRD response rate | through study completion,an average of 3 years
  To determine the Complete MRD response rate
Relapse rate | through study completion,an average of 3 years
  (time frame: at study completion, an average of 5 year)
Relapse-free survival | through study completion,an average of 3 years
  (time frame: at study completion, an average of 5 year)
Change in WT1 mRNA levels from peripheral blood samples and/or bone marrow biopsy samples. | through study completion,an average of 3 years
  Efficacy assessment will also be performed on a molecular level. Bone marrow biopsy samples obtained from participants will be examined, and part of samples will be analyzed by qRT-PCR for WT1 expression.

CONTACTS AND LOCATIONS:
Overall Officials: Liangding Hu, M.D., Study Director — the Fifth Medical Center the PLA General Hospital; Liangding Hu, M.D., Principal Investigator — the Fifth Medical Center the PLA General Hospital
Locations (1):
- Department of hematology, Beijing, Beijing Municipality, China